CLINICAL TRIAL: NCT04862182
Title: The Value of Intrapartum Ultrasound in Predicting Mode of Delivery
Brief Title: Intrapartum Ultrasound in Predicting Mode of Delivery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gamal Omar Abdel Ghany hussein, Principle investigator (Obgyn specialist), Cairo University
Other Study IDs: Intrapartum Ultrasound
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Ultrasound Therapy; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Trans-perineal ultrasound — Intrapartum trans-perineal ultrasound in predicting the mode of delivery.

SUMMARY:
Determine the value of intrapartum scan measurement(s) in predicting the mode of delivery.

DETAILED DESCRIPTION:
The assessment and management of progress of labour is based on subjective clinical findings. The diagnosis of delay in labour and decisions regarding the timing and / or type of intervention(s) rely on clinical abdominal examination and digital vaginal assessment of the degree of cervical dilatation, the position of the presenting part of the baby and its station in relation to the maternal pelvis . Several studies have demonstrated the inaccuracy and the lack of consistency in such assessment between different practitioners especially in certain malpositions, malpresentations or with excessive subcutaneous tissue oedema .

One of the important clinical parameters that is assessed in labour is the position of the fetal head. Precise knowledge of fetal occiput position in labour is essential because some malpositions, like a persistent occiput posterior position is associated with higher risk of operative delivery and maternal and perinatal morbidity. The correct determination of head position is crucial before attempting any operative vaginal delivery. Moreover, knowing the exact presentation is also of paramount importance. For example, the differentiation between a face and a brow presentation is important in clinical management particularly that the engaging diameters of the latter presentation are too big in a term baby for a safe vaginal birth to occur, Sonographic assessment of fetal head position is best performed by transabdominal imaging in axial and sagittal planes .

Another parameter that is important in evaluating the progress of labour is the fetal head station. The fetal head station is the level of the fetal head in the birth canal relative to the plane of the maternal ischial spines. Serial clinical assessments by digital vaginal examination give an indication of the progress in head decent throughout the labour process, Sonographic assessment of fetal head station is best performed by transperineal ultrasound in the midsagittal or axial plane .

Several authors reported that ultrasound examination is more accurate and reproducible than clinical examination in the diagnosis of fetal head position and station and in the prediction of arrest of labor . It has also been suggested that ultrasound examination has the potential to stratify women who have a spontaneous vaginal delivery from those who end up having an operative birth Furthermore, it has been demonstrated that it is feasible to rely on ultrasound to predict the outcome of a planned operative vaginal birth .

However, currently, there is no consensus regarding the best timing of intrapartum scanning, at least for some of these measurements. Similar there is no general agreement regarding which measurements should be obtained and how useful if some of these measurements are integrated into a prediction model together with demographic or other clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Full Term pregnancy
* Vertex presentation
* Singleton pregnancy
* In labour

Exclusion Criteria:

* Multiparous women
* Preterm labour
* Non vertex presentation
* Multi-fetal pregnancy
* Planned for elective Cesarean Section
* Underlying medical diseases
* Those unwilling to participate in the study

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Women who present to the labour ward in the first stage of labour and willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The rate of intrapartum Cesarean Section | 3 hours
  number of women that failed to progress to normal vaginal delivery and need for intrapartum Cesarean Section (ICS)

REFERENCES:
- [Result] Barak O, Levy R, Flidel O, Zaks S, Gillor M, Hagay Z, Vaisbuch E. The Routine Use of Intrapartum Ultrasound in Clinical Decision-Making during the Second Stage of Labor - Does It Have Any Impact on Delivery Outcomes? Gynecol Obstet Invest. 2018;83(1):9-14. doi: 10.1159/000455847. Epub 2017 Feb 22. PMID 28222431
- [Result] Brunelli E, Del Prete B, Casadio P, Pilu G, Youssef A. The dynamic change of the anteroposterior diameter of the levator hiatus under Valsalva maneuver at term and labor outcome. Neurourol Urodyn. 2020 Nov;39(8):2353-2360. doi: 10.1002/nau.24494. Epub 2020 Aug 31. PMID 32865824
- [Result] Sherer DM, Abulafia O. Intrapartum assessment of fetal head engagement: comparison between transvaginal digital and transabdominal ultrasound determinations. Ultrasound Obstet Gynecol. 2003 May;21(5):430-6. doi: 10.1002/uog.102. PMID 12768551
- [Result] Lipschuetz M, Cohen SM, Lewkowicz AA, Amsalem H, Haj Yahya R, Levitt L, Yagel S. [PROLONGED SECOND STAGE OF LABOR: CAUSES AND OUTCOMES]. Harefuah. 2018 Nov;157(11):685-690. Hebrew. PMID 30457229